CLINICAL TRIAL: NCT06372912
Title: Incidence of Early Postoperative Complications in Patients Undergoing Bariatric Surgery in 2022 Tijuana, Baja California
Brief Title: Early Postoperative Complications in Patients Undergoing Bariatric Surgery
Status: Recruiting | Type: Observational
Sponsor: Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Principal Investigator, GONZALEZ-OJEDA ALEJANDRO, Principal Investigator, Instituto Mexicano del Seguro Social
Other Study IDs: Complications-Bariatric-TJ
Record Dates: First submitted 2024-04-15; First posted 2024-04-18 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Bariatric Surgery Candidate; Complication,Postoperative
MeSH Terms: conditions — Postoperative Complications | interventions — Gastric Bypass

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing bariatric surgery
  Interventions: Procedure: Sleeve gastrectomy, Roux-en-Y gastric bypass, mini-gastric bypass, SADIS, intragastric balloon insertion, and gastric band placement are bariatric surgeries.

INTERVENTIONS:
Procedure: Sleeve gastrectomy, Roux-en-Y gastric bypass, mini-gastric bypass, SADIS, intragastric balloon insertion, and gastric band placement are bariatric surgeries. — Sleeve gastrectomy: reduces stomach size. Roux-en-Y gastric bypass: limits calorie absorption. Mini gastric bypass: achieves weight loss with fewer incisions. SADIS: combines sleeve gastrectomy with small bowel bypass. Intragastric balloon: reduces stomach volume. Gastric banding: restricts food intake.

SUMMARY:
This study examined immediate postoperative complications in patients undergoing various bariatric surgeries, aiming to evaluate the safety and efficacy of these interventions. Conducted at specialized high-volume bariatric surgery centers in Tijuana, Mexico. Predominantly female patients with severe obesity underwent procedures like sleeve gastrectomy and Roux-en-Y gastric bypass. Immediate complications were rare, occurring in only 0.38% of patients, with bleeding being the most common issue. Surgical reintervention within 48 hours was required in 0.33% of cases. The study's low complication rate suggests that surgeon expertise is crucial in minimizing risks and improving postoperative outcomes in bariatric surgery.

DETAILED DESCRIPTION:
This study, conducted in specialised high-volume bariatric surgery centres in Tijuana, Baja California, Mexico, aimed to analyze the outcomes of various bariatric surgery procedures. It include patients who underwent surgeries like sleeve gastrectomy, gastric bypass, and others. The surgeries were performed by five specialized surgeons with assistance from ten bariatric surgery subspecialists. The researchers reviewed electronic medical records and excluded patients with incomplete information. Postoperative complications requiring additional medical or surgical interventions were noted. Statistical analysis was conducted using SPSS software, focusing on descriptive measures like frequencies, percentages, means, and standard deviations.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and above
* Varying degrees of overweight or obesity who underwent surgery at the participating hospitals

Exclusion Criteria:

* incomplete or insufficient information in their medical records

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study included patients aged 18 and above with varying degrees of overweight or obesity who underwent bariatric surgery at specialized centers in Tijuana, Mexico. The surgeries examined were sleeve gastrectomy, Roux-en-Y gastric bypass, mini-gastric bypass, SADIS, intragastric balloon insertion, and gastric band placement. These procedures were performed by five bariatric surgery specialists with assistance from ten certified subspecialists. Patients with incomplete medical records were excluded. Immediate postoperative complications were defined as events requiring additional medical or surgical interventions beyond routine care.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of Postoperative Complications | 30 days
  Within 30 days following surgery, the incidence of anastomotic leaks and surgical site bleeding is the main safety consequence. This outcome measure is essential for proving the safety and enhanced recovery profile, since the technique emphasizes rigorous hemostasis and anastomotic integrity-achieved through reinforced suturing and patency verification using methylene blue tests.

SECONDARY OUTCOMES:
Long-term Weight Loss Efficacy | 12 months
  : The percentage of excess weight loss (%EWL) at 12 months after surgery is the main indicator of efficacy. One of the main objectives of bariatric surgery is to achieve significant and long-lasting weight loss. The percentage EWL is calculated using the patient's weight reduction from pre-surgery to a year after surgery, normalized to their excess weight using optimum body weight guidelines.

CONTACTS AND LOCATIONS:
Overall Officials: Jesús E Ortiz Gómez, MD, PhD, Study Director — Elias Ortiz & Company Mexico Weight Loss Specialists. Ernesto Sarmiento 2308, Tijuana 22046, Baja California, Mexico.; Almino Cardoso Ramos, MD, PhD, Study Chair — Elias Ortiz & Company Mexico Weight Loss Specialists. Ernesto Sarmiento 2308, Tijuana 22046, Baja California, Mexico.; Jaime Ponce de León Palomares, MD, PhD, Study Chair — Obesity Goodbye Center, Tijuana 2050, Baja California, Mexico.; José S Verboonen Sotelo, MD, PhD, Study Chair — Obesity Goodbye Center, Tijuana 2050, Baja California, Mexico; Jeffry Romero Manzano, MD, PhD, Study Chair — Obesity Goodbye Center, Tijuana 2050, Baja California, Mexico.; Isaac Esparza Estrada, MD, PhD, Study Chair — Obesity Goodbye Center, Tijuana 2050, Baja California, Mexico; Alejandro González Ojeda, MD, PhD, Study Chair — Professor at the Faculty of Medicine of the Universidad de Colima. Colima, Mexico; Christian Rodríguez López, MD, PhD, Study Chair — Body Art Surgical, Edificio Corporativo Central, Diego Rivera 2311, Zona Urbana Rio Tijuana, 22010 Tijuana, Baja California, Mexico.; Clotilde Fuentes-Orozco, MD, PhD, Study Chair — Senior Researcher B, Biomedical Research. Unidad de Investigación Biomédica 02, Unidad Médica de Alta Especialidad, Hospital de Especialidades del Centro Médico Nacional de Occidente del Instituto Mexicano del Seguro Social. Guadalajara, Jalisco. México; Sergio J Vázquez-Sánchez, MD, Study Chair — Unidad de Investigación Biomédica 02, Unidad Médica de Alta Especialidad, Hospital de Especialidades del Centro Médico Nacional de Occidente del Instituto Mexicano del Seguro Social; Hector J Pérez Corzo, MD, PhD, Study Chair — Renew Bariatrics, Bariatric Surgery Department, Tijuana, Baja California, Mexico; José O Orozco Álvarez Malo, MD, PhD, Study Chair — Colegio de Cirujanos Bariatras y Enfermedades Metabólicas del Estado de Baja California. Tijuana 2050, Baja California, Mexico.; Jhonattan A Barriga Fong, MD, PhD, Study Chair — Colegio de Cirujanos Bariatras y Enfermedades Metabólicas del Estado de Baja California. Tijuana 2050, Baja California, Mexico
Locations (1):
- Elias Ortiz & Company Mexico Weight Loss Specialists. Ernesto Sarmiento 2308, Tijuana 22046, Baja California, Mexico., Tijuana, Estado de Baja California, Mexico

IPD SHARING:
Plan to Share IPD: No